CLINICAL TRIAL: NCT01731275
Title: A Phase 1 Single Dose Study of E6011 in Japanese Healthy Adult Male Subjects
Brief Title: A Phase 1 Single Dose Study of E6011 in Japanese Healthy Adult Male Subjects (Study E6011-J081-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E6011-J081-001
Record Dates: First submitted 2012-08-31; First posted 2012-11-21 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Healthy Male Volunteers
Keywords: Healthy volunteers; immunogenicity; anti-E6011 antibody
MeSH Terms: interventions — quetmolimab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- E6011 (Experimental)
  Interventions: Drug: E6011
- E6011 Matching Placebo (Placebo Comparator)
  Interventions: Drug: E6011 Matching Placebo

INTERVENTIONS:
Drug: E6011 — A single ascending dose (SAD) administration of E6011 is administered to 8 groups as a 30-minute intravenous infusion at a dose of either 0.0006, 0.006, 0.04, 0.2, 1, 3, 6, or 10 mg/kg. Each participant in each group will receive a single-dose only once. The study drug will not be administered to more than two participants on the same day, and the second participant must start the study treatment after at least a 2-hour interval from the start of the study treatment in the first participant. The subsequent ascending dose groups will start approximately at least every 3 weeks following the study treatment in the first participant of each group.
  Arms: E6011
Drug: E6011 Matching Placebo — A SAD administration of E6011 Matching Placebo is administered to 2 participants in each of 8 groups as a 30-minute intravenous infusion at a placebo dose of either 0.0006, 0.006, 0.04, 0.2, 1, 3, 6, or 10 mg/kg. Each participant in each group will receive a single-dose only once. The study drug will not be administered to more than two participants on the same day, and the second participant must start the study treatment after at least a 2-hour interval from the start of the study treatment in the first participant. The subsequent ascending E6011 Matching Placebo dose groups will start approximately at least every 3 weeks following the study treatment in the first participant of each group.
  Arms: E6011 Matching Placebo

SUMMARY:
To evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of a single ascending dose (SAD) administration of E6011 in Japanese healthy volunteers.

ELIGIBILITY:
Inclusion criteria;

1. Non-smoking Japanese male subjects aged >= 20 to less than 45 years
2. BMI at screening is >= 18.5 kg/m2 to less than 25.0 kg/m^2
3. Males who have not had a successful vasectomy and their female partners must agree to practice highly effective contraception throughout the study period.

Exclusion criteria;

1. Has been treated with biologic products (except for immunoglobulin preparation)
2. Have received immunoglobulin or blood preparation within 6 months before the study drug administration
3. Received inoculation within 4 weeks before the study drug administration
4. Has a history of autoimmune disease or immunodeficiency
5. Has a clinically significant angioedema, hematemesis, anal hemorrhage, or hemoptysis
6. Has a history of acute myocardial infarction, cerebral infarction, cerebral hemorrhage, or arteriosclerosis obliterate
7. With gross hematuria, occult bleeding in urine (>=1+) and urine protein (>=1+) , or either of (>=2+) at screening
8. Has a clinically significant vasculitis (e.g., multiple mononeuropathy)
9. Known to be positive for human immunodeficiency virus (HIV antigen and antibody), hepatitis B virus surface antigen (HBs antigen), hepatitis B virus surface antibody (HBs antibody), hepatitis B virus (HBV) DNA, hepatitis C virus (HCV) antibody, or syphilis serology test
10. Known to be positive for human T-cell lymphotropic virus type 1 (HTVL-1) antibody at screening
11. Known to be positive for QuantiFERON-TB Gold Test
12. Treated with ethical drug(s) within 4 weeks before the study drug administration (except for disinfectants, eye drops)
13. Treated with non-prescription drug(s) within 2 weeks before the study drug administration (except for disinfectants, eye drops)
14. Has participated in another clinical trial and received an investigational drug or device within 6 months before the study drug administration
15. Received blood transfusion within 1 year, 400 mL or more whole blood donation within 12 weeks, or 200 mL or more whole blood donation within 4 weeks, or blood constituent donation within 2 weeks before the study drug administration.

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Up to Week 24
  An Adverse Event (AE) is any untoward medical occurrence in a participant administered an investigational product. An AE does not necessarily have a causal relationship with the medicinal product. The investigator or sub-investigator reviews all laboratory findings and determines if they constitute an AE. In-patient observation assessments will be performed during 1 week post-dose, followed by the out-patient observation assessments in groups: 0.0006, 0.006, 0.04, 0.2 mg/kg up to the end of Week 8 and in groups: 1, 3, 6, 10 kg/mg) up to the end of Week 24.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Up to 24 Weeks post-dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Up to 24 Weeks post-dose
Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] | Up to 24 Weeks post-dose
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t).
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - infinity)] | Up to 24 Weeks post-dose
  AUC (0 - infinity)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - infinity). It is obtained from AUC (0 - t) plus AUC (t - infinity).
Plasma Decay Half-Life (t1/2) | Up to 24 Weeks post-dose
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Pharmacokinetic Parameter: Volume of Distribution (Vd) | Up to 24 Weeks post-dose
Pharmacokinetic Parameter: Clearance (CL) | Up to 24 Weeks post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Kiyoshi Oketani, Study Director — KAN Clinical Development Section, JAPAN/ASIA Clinical Research Product Creation Unit, Eisai Product Creation System
Locations (1):
- Sagamihara, Kanagawa, Japan